CLINICAL TRIAL: NCT04299607
Title: Performance Assessment of the DPP Fever Panel II Assay for Detection of Infectious Causes of Acute Febrile Illness in Laos
Brief Title: Evaluation of the DPP II Assay in Laos
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: FE004
Record Dates: First submitted 2019-11-26; First posted 2020-03-09 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Acute Febrile Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AFI patients: Blood will be collected from patients presenting with an undifferentiated fever.
  Samples will be tested with:
  * the Malaria Ag Pf/Pan test SD Bioline
  * the SD Bioline Dengue Duo IgM/IgG/NS1
  * the DPP Zika Chikungunya Dengue test from Chembio
  * the DPP Fever Panel II assay
  * the Leptospira IgM ELISA test from Serion
  * an in-house ELISA tests for scrub and murine typhus IgM
  * blood culture for detection of Burkholderia pseudomallei
  Interventions: Diagnostic Test: DPP Fever Panel II assay and DPP Micro Readers

INTERVENTIONS:
Diagnostic Test: DPP Fever Panel II assay and DPP Micro Readers — Detection of common causes of acute febrile illnesses in Asia

SUMMARY:
Fever is the most frequent symptom in patients seeking care globally. Several causative agents of febrile illness have been described with a high prevalence in South East Asia. They include malaria, dengue, Rickettsia, Leptospira and Burkholderia species. Since their introduction in the market, rapid diagnostic tests for malaria have driven patient management and care. Malaria negative cases are commonly treated with antibiotics without confirmation of bacteraemia. This can be explained by conventional laboratory diagnostic tests such as blood culture that usually require a skilled staff and appropriate facilities.

Several Rapid Diagnostic tests (RDTs) are currently in the market but only limited data on their performance are available, rendering them unsuitable to replace laboratory conventional tests. In addition, RDTs have been developed for single disease diagnosis and remain costly for Low and Middle Income Countries (LMIC).

Chembio, in collaboration with FIND (Foundation for Innovative New Diagnostics) and MORU (Mahidol Oxford Tropical Medicine Research Unit), has developed a multiplex lateral flow immunoassay (DPP® Fever Panel II Assay) that is able to detect serum immunoglobulin M (IgM) and specific microbial antigen of the most common agents of Acute Febrile Illness (AFI) in Asia. The assay comes with a reader that provides results interpretation to the operator.

So far, DPP II assay performance has been estimated using a limited number of retrospective serum samples. More data are required to assess the performance of the assay using prospective serum samples. In addition, only limited data are available regarding the performance of the assay using blood samples. FIND will conduct a clinical trial to estimate the clinical performance of the assay in comparison to reference tests, using blood and serum samples and in intended settings of use.

ELIGIBILITY:
Inclusion Criteria:

* Participants > 12 years old enrolled in the "Prospective study of the causes of fever amongst patients admitted to Mahosot Hospital, Vientiane, Lao PDR" (UI-2 study).
* Fever (≥ 37.5 °C)
* Illness duration < 14 days
* Willingness to provide blood samples by venepuncture

Exclusion Criteria:

* Absence of consent (and assent for children) to participate to the "Prospective study of the causes of fever amongst patients admitted to Mahosot Hospital, Vientiane, Lao PDR" (UI-2 study).
* Non-infectious known or suspected cause of fever
* No left over blood sample or insufficient volume of left over sample

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population consists of samples collected from individuals who consent to participate to the "Prospective study of the causes of fever ("UI-2" Study) amongst patients admitted to Mahosot Hospital, Vientiane, Lao PDR" (OxTREC reference: 006-07). Individuals provide blood samples for routine laboratory tests and blood leftovers will be used during this trial.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Percentage of samples with concordant results for marker detection in paired whole blood and serum samples for each reader | 5 months
  The percentage of samples with concordant results using two types of assay readers will be calculated for each marker and each specimen type (blood and serum)
Optimal reader cut-offs for serum samples and for blood samples to obtain the overall highest diagnostic accuracy per sample type | 5 months
  The reader cut-offs (numerical values) that give the highest specificity and specificity will calculated for each marker and reader
Percentage of more targeted treatments that would have been prescribed if the DPP II assay test was used in routine in comparison to actual prescribed treatments and to treatment that would have been prescribed based on comparator tests | 5 months
  In comparison to reference tests and routine tests, the impact of the DPP Fever Panel II assay on antibiotic prescriptions will be modeled
Cost impact of more targeted treatments that would have been prescribed if the DPP II assay test was used in routine in comparison to actual prescribed treatments and to treatment that would have been prescribed based on comparator tests | 5 months
  In comparison to reference tests and routine tests, the impact of the DPP Fever Panel II assay on health costs will be modeled.

SECONDARY OUTCOMES:
Estimates of sensitivity and specificity of the DPP assay for detection of fever causative agents using venous blood samples, in comparison to reference tests | 5 months
Estimates of sensitivity and specificity of the DPP assay for detection of fever causative agents using serum samples, in comparison to reference tests. | 5 months
Estimates of operational characteristics, including invalid and indeterminate rates | 5 months
  The % of invalid results and indeterminate rates will be calculated.
Estimates of ease-of-use will be captured through user-appraisal questionnaire. | 5 months
  Answers to each question will be graded either positive, neutral or negative. The % and absolute numbers of positive, neutral and negative answers will be reported in tables and charts.

CONTACTS AND LOCATIONS:
Locations (1):
- LOMWRU, Mahosot Hospital, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: Undecided